CLINICAL TRIAL: NCT01209208
Title: Double-blind, Double-dummy, Randomised, Placebo-controlled, Multi-centre Phase III Study on the Efficacy and Tolerability of a 8-week Treatment With Budesonide vs. Mesalazine vs. Placebo in Patients With Lymphocytic Colitis
Brief Title: Budesonide Versus Mesalazine Versus Placebo in Lymphocytic Colitis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Dr. Falk Pharma GmbH (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: BUG-1/LMC; 2008-005994-36 (EudraCT Number)
Record Dates: First submitted 2010-09-23; First posted 2010-09-27 (Estimated); Last update posted 2017-07-26 (Actual); Status verified 2017-07

CONDITIONS: Lymphocytic Colitis
MeSH Terms: conditions — Colitis, Lymphocytic | interventions — Budesonide; Mesalamine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- A (Experimental): Budesonide
  Interventions: Drug: Budesonide
- B (Experimental): Mesalazine
  Interventions: Drug: Mesalamine
- C (Placebo Comparator)
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Budesonide — 9 mg per day
  Arms: A
Drug: Mesalamine — 3 g per day
  Arms: B
Other: Placebo — 0 g per day
  Arms: C

SUMMARY:
The purpose of this study is to determine whether budesonide or mesalazine is more active in the treatment of lymphocytic colitis.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent
* Symptoms and signs of indication of lymphocytic colitis

Exclusion Criteria:

* Infectious diarrhoea,
* Diarrhoea as a result of the presence of other symptomatic organic disease(s) of the gastrointestinal tract or endoscopic-histological findings Celiac disease
* Pregnancy or breast-feeding,
* Participation in an other clinical trial

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 57 (Actual)
Dates: Start 2010-05; Primary Completion 2017-06 (Actual); Study Completion 2017-06 (Actual)

PRIMARY OUTCOMES:
Rate of clinical remission | 8 weeks

SECONDARY OUTCOMES:
Proportion of patients with histological improvement | 8 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Stephan Miehlke, Professor, Principal Investigator — Magen-Darm-Zentrum, IKE - Internistische Kooperation Eppendorf, Hamburg, Germany
Locations (1):
- Magen-Darm-Zentrum, IKE - Internistische Kooperation Eppendorf, Hamburg, Germany

REFERENCES:
- [Derived] Miehlke S, Aust D, Mihaly E, Armerding P, Bohm G, Bonderup O, Fernandez-Banares F, Kupcinskas J, Munck LK, Rehbehn KU, Nacak T, Greinwald R, Munch A; BUG-1/LMC Study Group. Efficacy and Safety of Budesonide, vs Mesalazine or Placebo, as Induction Therapy for Lymphocytic Colitis. Gastroenterology. 2018 Dec;155(6):1795-1804.e3. doi: 10.1053/j.gastro.2018.08.042. Epub 2018 Sep 7. PMID 30195447